CLINICAL TRIAL: NCT02865382
Title: Detection of Colorectal Adenoma by Optical Enhancement Technology vs. High-Definition Colonoscopy: A Randomized Trial
Brief Title: Detection of Colorectal Adenoma by Optical Enhancement Technology vs. High-Definition Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, Professor, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2016SDU-QILU-11
Record Dates: First submitted 2016-08-02; First posted 2016-08-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-08

CONDITIONS: Colonic Polyps
Keywords: Adenoma detection rate; Optical Enhancement Technonogy; Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): white light was used for both insertion and withdrawal of the colonoscope
  Interventions: Procedure: white light was used for colonoscopy withdrawal
- Group B (Experimental): Insertion to cecum was performed under white light and once the cecum was reached,the OE mode was swithed on during withdrawal of endoscope for complete colonic examination
  Interventions: Procedure: OE mode was used for colonoscopy withdrawal

INTERVENTIONS:
Procedure: white light was used for colonoscopy withdrawal
  Arms: Group A
Procedure: OE mode was used for colonoscopy withdrawal
  Arms: Group B

SUMMARY:
Optical Enhancement Technology might be superior to the conventional HD-WL in detecting colorectal adenomas

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer in the world.Colonoscopy is the gold standard screening test for colorectal cancer.There are also emerging data to support that screening by colonoscopy reduces both the incidence and mortality of colorectal cancer.However,Colonoscopy could still miss colorectal adenomas and even cancer.The miss rate for colonic adenomas was reported to be ranging from 15 to 32% in tandem colonoscopy studies.The reasons for the miss rate may be technical(insufficient during excessively fast instrument withdrawal),but may also be the imaging method.Smaller lesions ,particularly flat ones ,may be missed as a result of their subtle appearance and limited contrast in relation to the surrounding mucosa.

Some image-enhanced modules were developed with an aim to improve colorectal polyp or adenoma detection.The widely available modules is the narrow band imaging(NBI).However,most studies failed to demonstrate any superiority of NBI system over white light colonoscopy in detecting colonic polyps.NBI provides dimmer images of the colonic mucosa ,which may limit its performance on polyp and adenoma detection.

Like NBI,OE technology is image-enhanced module,providing a more intense look at the vascular pattern morphology.Besides,OE technology provides an much brighter image compared to NBI.This may possibly increase polyp detection by enhancing visibility of the colonic mucosa with brighter image.The current study aims to tested whether OE technology would improve adenoma detection when compared with high-definition colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients were selected if they presented for diagnostic colonoscopy for a variety of indications(eg positive fecal occult blood test, abdominal pain, diarrhoea,post-polypectomy surveillance).

Exclusion Criteria:

* Patients with prior resection of the proximal colon, advanced colonic cancer, inflammatory bowel disease, or polyposis syndrome.
* The cecum could not be intubated.
* Inadequate bowel preparation (Aronchick Bowel Preparation Scale score poor or inadequate).
* Biopsies were not available.
* Unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
adenoma detection rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD, PhD, Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong Province, China
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Adler A, Pohl H, Papanikolaou IS, Abou-Rebyeh H, Schachschal G, Veltzke-Schlieker W, Khalifa AC, Setka E, Koch M, Wiedenmann B, Rosch T. A prospective randomised study on narrow-band imaging versus conventional colonoscopy for adenoma detection: does narrow-band imaging induce a learning effect? Gut. 2008 Jan;57(1):59-64. doi: 10.1136/gut.2007.123539. Epub 2007 Aug 6. PMID 17681999
- [Background] Aminalai A, Rosch T, Aschenbeck J, Mayr M, Drossel R, Schroder A, Scheel M, Treytnar D, Gauger U, Stange G, Simon F, Adler A. Live image processing does not increase adenoma detection rate during colonoscopy: a randomized comparison between FICE and conventional imaging (Berlin Colonoscopy Project 5, BECOP-5). Am J Gastroenterol. 2010 Nov;105(11):2383-8. doi: 10.1038/ajg.2010.273. Epub 2010 Jul 13. PMID 20628363